CLINICAL TRIAL: NCT04871906
Title: The Effect of Stretching Exercises on Vascular Function, Blood Flow, and Walking Function in Middle and Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Mei-Wun Tsai, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: YM109100E
Record Dates: First submitted 2021-04-26; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Stretch
Keywords: stretching exercise; vascular function; blood flow; walking function; fitness
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching exercises (Experimental): Interventions are home-based stretching exercises. The experimental group will receive 6 stretching exercises which stretch 20-30 seconds, relax for 10 seconds, and repeat 5 times for each side. It will take 25-30 minutes every day for continuous 8 weeks.
  Interventions: Other: stretching exercises
- Control group (No Intervention): Maintain their daily activity level in the 8 weeks. We use the study desigh-''waiting list control'' in this group.

INTERVENTIONS:
Other: stretching exercises — Our interventions are home-based stretching exercises. The experimental group will receive 6 stretching exercises which stretch 20-30 seconds, relax for 10 seconds, and repeat 5 times for each side. It will take 25-30 minutes every day for continuous 8 weeks. Those include stretching of the deep front line, spiral line, superficial front line, lateral line, superficial back line, and plantar flexors. Designed concepts are the following three: 1) based on ''Anatomy- Train'' theory, 2) emphasize on movements of trunk and pelvis, and 3) stress on the stretching of lower extremities.
  Arms: Stretching exercises

SUMMARY:
This study examines the relationship between circulation and walking speed after performing 8-week stretching exercises.

DETAILED DESCRIPTION:
This study examines the relationship between circulations and walking speeds. Most studies in the field of stretching exercises have only focused on improvements of endothelial functions in younger population; however, I aim to emphasize its effects on different populations, such as people with frailty, low physical activity level, weakness and postoperative status. Previous research has established that stretching exercises can improve walking function by modulations of musculoskeletal or neuromuscular system. The importance and originality of this study are that it explores the relationship between circulation and walking speed. Due to the inability to extrapolate outcomes; short-term effect of improved blood vessel function; the unclear mechanism of stretching exercises; and considering the different physical fitness groups, I design a home-based, low-dose, and anatomic chain-based stretching exercises to verify the possible mechanism and effects.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20-85 years old
2. Follow instructions
3. Walk with/without assistive technology

Exclusion Criteria:

1. Unstable acute or chronic health conditions
2. Peripheral vascular diseases
3. Non-musculoskeletal problems that would limit stretching exercises
4. Participate in other exercise programs

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
vascular functions-Stiffness index(1) | pre-intervention(1st week)
  (Stiffness index, SI，unit：m/s)
vascular functions-Stiffness index(2) | during intervention(4th week)
  (Stiffness index, SI，unit：m/s)
vascular functions-Stiffness index(3) | post-intervention(8th week)
  (Stiffness index, SI，unit：m/s)
vascular functions-Reflective index(1) | pre-intervention(1st week)
  (Reflective index, RI，unit：％)
vascular functions-Reflective index(2) | during intervention(4th week)
  (Reflective index, RI，unit：％)
vascular functions-Reflective index(3) | post-intervention(8th week)
  (Reflective index, RI，unit：％)
vascular functions-Vascular age | pre-intervention(1st week)
  (Vascular age, VA，unit：year-old)
Ultrasound parameters-peak-systolic velocity(1) | pre-intervention(1st week)
  （peak-systolic velocity, PSV)
Ultrasound parameters-peak-systolic velocity(2) | during intervention(4th week)
  （peak-systolic velocity, PSV）
Ultrasound parameters-peak-systolic velocity(3) | post-intervention(8th week)
  （peak-systolic velocity, PSV）
Ultrasound parameters-end-diastolic velocity(1) | pre-intervention(1st week)
  （end-diastolic velocity, EDV）
Ultrasound parameters-end-diastolic velocity(2) | during intervention(4th week)
  （end-diastolic velocity, EDV）
Ultrasound parameters-end-diastolic velocity(3) | post-intervention(8th week)
  （end-diastolic velocity, EDV）
Ultrasound parameters-mean velocity(1) | pre-intervention(1st week)
  （mean velocity, mV）
Ultrasound parameters-mean velocity(2) | during intervention(4th week)
  （mean velocity, mV）
Ultrasound parameters-mean velocity(3) | post-intervention(8th week)
  （mean velocity, mV）
Ultrasound parameters-mean volume flow(1) | pre-intervention(1st week)
  (mean volume flow, vFl)
Ultrasound parameters-mean volume flow(2) | during intervention(4th week)
  (mean volume flow, vFl)
Ultrasound parameters-mean volume flow(3) | post-intervention(8th week)
  (mean volume flow, vFl)
Ultrasound parameters-resistance index(1) | pre-intervention(1st week)
  (resistance index, RI)
Ultrasound parameters-resistance index(2) | during intervention(4th week)
  (resistance index, RI)
Ultrasound parameters-resistance index(3) | post-intervention(8th week)
  (resistance index, RI)
Ultrasound parameters-pulsatility index(1) | pre-intervention(1st week)
  (pulsatility index, PI)
Ultrasound parameters-pulsatility index(2) | during intervention(4th week)
  (pulsatility index, PI)
Ultrasound parameters-pulsatility index(3) | post-intervention(8th week)
  (pulsatility index, PI)
Ultrasound parameters-diameter(1) | pre-intervention(1st week)
  （diameter, D）
Ultrasound parameters-diameter(2) | during intervention(4th week)
  （diameter, D）
Ultrasound parameters-diameter(3) | post-intervention(8th week)
  （diameter, D）
Ultrasound parameters-area(1) | pre-intervention(1st week)
  （area, A）
Ultrasound parameters-area(2) | during intervention(4th week)
  （area, A）
Ultrasound parameters-area(3) | post-intervention(8th week)
  （area, A）
walking speed-preferred(1) | pre-intervention(1st week)
  Timed 10-Meter Walk Test (preferred)
walking speed-preferred(2) | during intervention(4th week)
  Timed 10-Meter Walk Test (preferred)
walking speed-preferred(3) | post-intervention(8th week)
  Timed 10-Meter Walk Test (preferred)
walking speed-fast(1) | pre-intervention(1st week)
  Timed 10-Meter Walk Test (fast)
walking speed-fast(2) | during intervention(4th week)
  Timed 10-Meter Walk Test (fast)
walking speed-fast(3) | post-intervention(8th week)
  Timed 10-Meter Walk Test (fast)

SECONDARY OUTCOMES:
body composition-height | pre-intervention(1st week)
  height(cm)
body composition-weight | pre-intervention(1st week)
  weight(kg)
body composition-waist circumference | pre-intervention(1st week)
  waist circumference(cm)
vital sign-blood pressure(1) | pre-intervention(1st week)
  blood pressure(mmHg)
vital sign-blood pressure(2) | during intervention(4th week)
  blood pressure(mmHg)
vital sign-blood pressure(3) | post-intervention(8th week)
  blood pressure(mmHg)
vital sign-heart rate(1) | pre-intervention(1st week)
  heart rate(bpm)
vital sign-heart rate(2) | during intervention(4th week)
  heart rate(bpm)
vital sign-heart rate(3) | post-intervention(8th week)
  heart rate(bpm)
flexibility-chair sit and reach test (1) | pre-intervention(1st week)
  chair sit and reach test (cm)
flexibility-chair sit and reach test (2) | during intervention(4th week)
  chair sit and reach test (cm)
flexibility-chair sit and reach test (3) | post-intervention(8th week)
  chair sit and reach test (cm)
grip strength | pre-intervention(1st week)
  hand dynamometer
cognitive function | pre-intervention(1st week)
  Montreal Cognitive Assessment.Minimum value is 0 and maximum value is 30, and higher scores mean a better outcome
frailty | pre-intervention(1st week)
  SOF (Study of Osteoporotic Fractures). Minimum value is 0 and maximum value is 3, and higher scores mean a worse outcome
basic data | pre-intervention(1st week)
  gender, age, education, living status, smoking, and exercise habits
ACSM-PAR-Q+ | pre-intervention(1st week)
  The Physical Activity Readiness Questionnaire for Everyone AND follow-up questions about their medical conditions (PAR-Q+) is used to identify whether subjects are at risk in engaging in exercises. Thus, researchers can prescribe individual exercise prescriptions.
IPAQ | pre-intervention(1st week)
  International Physical Activity Questionnaire to investigate their physical activity levels. Higher the amount of physical activity (min-METs/week) means a more active life-style(physical activity level).
fitness | pre-intervention(1st week)
  (Duke activity status index, DASI) Minimum value is 0 and maximum value is 58.2, and higher scores mean a better physical activity level.
adherence of exercise | post-intervention(8th week)
  usage records from the Line app

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Ying Lai, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan